CLINICAL TRIAL: NCT01372176
Title: Early Goal-Directed Nutrition in ICU Patients - EAT-ICU Trial
Acronym: EAT-ICU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other); Fresenius Kabi (Industry); European Society for Clinical Nutrition and Metabolism (Other)
Responsible Party: Principal Investigator, Matilde Jo Allingstrup, PhD Fellow, MSc Clinical Nutrition, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2011-002547-94
Record Dates: First submitted 2011-06-06; First posted 2011-06-13 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Critical Illness; Intensive Care (ICU) Myopathy; Muscle Wasting; Loss of Physical Function; Mechanical Ventilation
Keywords: Intensive care unit; Critical illness; Mortality; Reduced quality of life; Loss of lean body mass; Loss of physical function; Optimised nutritional support; Early initiation of nutrition; Indirect calorimetry
MeSH Terms: conditions — Critical Illness; Muscular Diseases; Muscular Atrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Goal-Directed Nutrition (Experimental)
  Interventions: Other: Early Goal-Directed Nutrition
- ASPEN-guidelines (Active Comparator)
  Interventions: Other: ASPEN-guidelines

INTERVENTIONS:
Other: Early Goal-Directed Nutrition — 1. Initiation of early supplementary parenteral nutrition (≤ 24 hours of admission).
  2. Measurement of requirements (indirect calorimetry, 24-hour urinary urea) leading to patient-specific, individualised and goal-directed nutritional therapy.
  3. Intervention goal: delivering 100% of patient-specific requirements, measured or calculated throughout entire admission (EN+PN).
  Arms: Early Goal-Directed Nutrition
Other: ASPEN-guidelines — EN will be the preferred route of nutrition, and will be initiated within the first 24 hours of ICU admission, in accordance with best evidence. The amount is gradually increased over the first days of admission as tolerated by the patient (assessed from gastric aspirates). If EN fails to reach calculated goals at day 7, supplementary PN will be initiated at admission day 8 to reach goals. Protein and energy goals will be calculated as 25 kcal/kg/day and 1.2 g protein/kg/day.
  Arms: ASPEN-guidelines

SUMMARY:
An increasing number of patients survive critical illness and intensive care, but describe having impaired physical function several years after discharge as a consequence of extensive loss of muscle mass. Reasons for loss of muscle mass and physical function are multiple, but insufficient nutrition is likely to contribute.

This randomised trial will investigate the effect of an optimised nutrition therapy during intensive care, on short term clinical outcome and physical quality of life. We hypothesise, that early nutritional therapy, directed towards patient-specific goals for energy and protein requirements, will improve both short- and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Acutely admitted to the ICU
* Expected length of stay in ICU > 3 days
* Mechanically ventilated, which enables indirect calorimetry
* Have central venous catheter wherein TPN can be administered
* Written proxy consent obtained (proxy consent defined as consent from two doctors, who are independent of the trial)
* Must be able to understand Danish

Exclusion Criteria:

* Contraindications to use enteral nutrition
* Contraindications to use parenteral nutrition, eg. hypersensitivity towards fish-, egg or peanut protein, or any of the active substances in the PN products
* Receiving a special diet
* Burns > 10% total body surface area
* Severe hepatic failure (Child-Pugh class C) or severe hepatic dysfunction: Bilirubin ≥ 50 µmol/l (3 mg/dl) + alanine aminotransferase ≥ 3 times upper reference value
* Traumatic brain injury
* Diabetic ketoacidosis
* Hyperosmolar non-ketotic acidosis
* Known or suspected hyperlipidemia
* BMI below 17 or severe malnutrition
* Pregnancy
* The clinician finds that the patient is too deranged (circulation, respiration, electrolytes etc.) or that death is imminent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2013-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Physical function | 6 months after randomisation
  Physical function 6 months after randomisation (physical component summary (PCS)-score of SF-36, conducted as phone-interview by a person blinded to the intervention

SECONDARY OUTCOMES:
Mortality | 28 days
Mortality | 90 days
Mortality | 6 months
Survival status for all patients | 6 months
New organ failure in the ICU | Followed until ICU discharge, an expected average of 21 days
  SOFA score above 3 in every category ex. Glasgow Coma Scale Score
Metabolic control | Followed until ICU discharge, an expected average of 21 days
  Accumulated insulin administration to maintain B-glucose ≤10 mmol/l and rates of severe hyper- and hypoglycaemia (B-glucose >15 mmol/l or ≤2.2 mmol/l, respectively)
New onset of renal replacement therapy | Followed until ICU discharge, an expected average of 21 days
Accumulated energy- and protein balance | Followed until ICU discharge, an expected average of 21 days
Length of stay in ICU | Up to 52 weeks
  Among survivors
Length of stay in hospital | Up to 52 weeks
  Among survivors
Serious adverse reactions in ICU | Up to 52 weeks
  Severe allergic reactions or elevated levels of liver enzymes in plasma
Health related quality of life | 6 months after randomisation
  Assessed by SF-36 questionnaire
Rate of nosocomial infections | Followed until ICU discharge, an expected average of 21 days
  Defined in six subcategories by a person blinded for the intervention
Percent days alive without inotropic/vasopressor support at day 90 | Up to 90 days
Percent days alive without renal replacement therapy at day 90 | Up to 90 days
Percent days alive without mechanical ventilation at day 90 | Up to 90 days
Cost analyses | Up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anders Perner, Professor, MD, PhD, Principal Investigator — Rigshospitalet, Department of Intensive Care; Matilde Jo Allingstrup, PhD Fellow, MSc, Study Director — Rigshospitalet, Department of Intensive Care
Locations (1):
- Department of Intensive Care, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Allingstrup MJ, Kondrup J, Wiis J, Claudius C, Pedersen UG, Hein-Rasmussen R, Bjerregaard MR, Steensen M, Jensen TH, Lange T, Madsen MB, Moller MH, Perner A. Early goal-directed nutrition versus standard of care in adult intensive care patients: the single-centre, randomised, outcome assessor-blinded EAT-ICU trial. Intensive Care Med. 2017 Nov;43(11):1637-1647. doi: 10.1007/s00134-017-4880-3. Epub 2017 Sep 22. PMID 28936712
- [Derived] Allingstrup MJ, Kondrup J, Wiis J, Claudius C, Pedersen UG, Hein-Rasmussen R, Jensen TH, Lange T, Perner A. Early goal-directed nutrition in ICU patients (EAT-ICU): protocol for a randomised trial. Dan Med J. 2016 Sep;63(9):A5271. PMID 27585532